CLINICAL TRIAL: NCT04174131
Title: A Prospective, Split-face, Randomized, Comparative Trial on the Efficacy of Two Hyaluronic Acid Products (Restylane + Lidocaine and Restylane Lyft) for the Treatment of Nasolabial Folds
Brief Title: Restylane + Lidocaine and Restylane Lyft for the Treatment of Nasolabial Folds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-Gal-004NLF
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Wrinkles Such as Nasolabial Folds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (right) B (left) (Experimental): Subjects will receive Restylane + Lidocaine and Restylane Lyft. One product will be randomized, per NLF.
  Interventions: Device: Restylane + Lidocaine; Device: Restylane® Lyft
- Treatment B (right) A (left) (Experimental): Subjects will receive Restylane + Lidocaine and Restylane Lyft. One product will be randomized, per NLF.
  Interventions: Device: Restylane + Lidocaine; Device: Restylane® Lyft

INTERVENTIONS:
Device: Restylane + Lidocaine — Restylane + Lidocaine is a HA gel generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL with 0.3% lidocaine. It is indicated for mid-to-deep dermal implantation for the correction of moderate to severe facial wrinkles and folds, such as NLFs.
Device: Restylane® Lyft — Restylane® Lyft is a sterile gel of HA with lidocaine generated by Streptococcus species of bacteria, chemically cross-linked with BDDE (the cross linker), stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL. Lyft is intended to be used for facial tissue augmentation (Galderma Laboratories, 2014).

SUMMARY:
This study is designed to assess and compare the efficacy of two hyaluronic acid (HA) fillers on moderate, severe and extreme nasolabial folds (NLF).

DETAILED DESCRIPTION:
Background

One of the most significant signs of aging is the appearance of deep lines that run from each side of the nose to the corners of the mouth [i.e., nasolabial folds (NLFs)]. These folds are defined by facial structures that support the buccal fat pad and separate the cheeks from the upper lip. The NLFs form due to volume shifts in the face, caused by a combination of fat descent and bone absorption, which results in sagging skin and hollowing.

Soft tissue augmentation can effectively restore the youthful, harmonious contours of the face. The most popular non-invasive treatment options for volume loss in the face include the use of hyaluronic acid (HA) fillers. Injections of HA for skin rejuvenation are one of the most common aesthetic treatments performed worldwide. Due to their effectiveness, safety, low immunogenicity (HA is a normal component of human skin) and reversibility with hyaluronidase, HA fillers are understandably a popular option for facial volume restoration.

Through recent advances in manufacturing technology, various types of HA fillers have been approved for the correction of facial wrinkles and folds, such as NLFs. Two such fillers, i) Restylane + Lidocaine and ii) Restylane Lyft, are well tolerated and provide significant improvement in this indication. These products contain the same amount of HA (i.e., 20mg/mL) and are manufactured using the same technology [i.e., non-animal stabilized hyaluronic acid (NASHATM)], but differ primarily in their particle size.

Small particle size HA (Restylane + Lidocaine): was the first non-animal stabilized HA-containing filler approved for use in the United States. Because of its particle size (i.e., 330-430 μM), Restylane + Lidocaine is referred to as small gel-particle HA (SGP-HA). NASHA small gel contains approximately 100,000 gel particles per mL.

Large particle size HA (Restylane Lyft): was approved in the United States in 2010 and is considered a large gel particle hyaluronic acid (LGP-HA). Restylane Lyft also contains the anesthetic lidocaine. NASHA large gel contains approximately 10,000 gel particles per mL.

The difference in gel size between the two products results in different viscosity and lifting capabilities, which is anticipated to affect treatment outcomes. While the comparative research is limited, a small number of clinical trials have compared the two products. For example, two randomized studies performed using US populations have shown equivalent safety and similar efficacy of Restylane + Lidocaine and Restylane Lyft, in subjects of all Fitzpatrick skin types; and one recent study found that both products exhibit similar safety and efficacy in a Chinese population. These three comparative studies found no significant differences in safety of LGP- and SGP-HA however, efficacy changes can occur due to the injection techniques and depth of injection used by the investigators.

This study is designed to assess and compare the efficacy of these two HA fillers on moderate, severe and extreme NLF, when using a modified technique. This modified technique will use a single puncture technique in each NLF, in comparison to others who have used a multi puncture, fanning or linear threading injection technique. For each NLF, a single bolus of product will be placed within the nasal pyriform aperture, on the periosteum. The location of the puncture will also vary from previous trials, in which injections were performed directly within the NLFs (to replace soft tissue volume). It is hypothesized that when these two products are used for replacing bone loss due to age-related resorption in the pyriform aperture, differences in efficacy will be observed that are not evident when they are used in soft tissue for volume augmentation. It is expected that while aesthetic outcomes and longevity of effect may be similar between the two products, the volumes required to achieve these same results will differ significantly, due to their different particle sizes.

Study Rationale

Larger HA gel particles result in better lifting capacities. Therefore, Restylane Lyft should display better efficacy in comparison to Restylane + Lidocaine when a "firm" product with a high lift capacity is required, such as when trying to replace or reshape bone. This is in contrast to replacing soft tissue volume, which was evaluated in earlier studies. However, as previous authors have reported, when these two products are used to replace soft tissue volume they both provide adequate lifting capabilities and thus result in similar efficacy levels.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, women between the ages of 30 and 75 years old;
2. Indication for treatment of bilateral NLFs and wrinkles;
3. Willingness to comply with study requirements;
4. Provide written consent;
5. Accepted the obligation not to receive any other facial procedures through the follow-up;
6. Understood and accepted the obligation and would be logistically able to appear for all scheduled follow-up visits;
7. No previous facial fillers for a period of 12 months prior to this study;
8. No previous facial fillers in the complete region of the NLF for 18 months prior to this study

Exclusion Criteria:

1. Current pregnancy or lactation [sexually active women of childbearing age must agree to use medically acceptable methods of contraception for the duration of this study (e.g., oral contraceptives, condoms, intrauterine device, shot/injection, patch)];
2. Hypersensitivity to hyaluronic acid or local anesthetics;
3. Patients meeting any official Restylane contra-indications;
4. Patients presenting with porphyria;
5. Inability to comply with follow-up and abstain from facial injections during the study period;
6. Heavy smokers, classified as smoking more than 12 cigarettes per day;
7. History of severe or multiple allergies manifested by anaphylaxis;
8. Previous tissue revitalization therapy in the treatment area within 6 months before treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling, or dermabrasion;
9. Previous maxillofacial surgery including aesthetic facial surgical therapy or liposuction, piercing, or tattoos in the treatment area;
10. History or presence of any disease or lesion near or at the treatment area, including inflammation, active or chronic infection, including in the mouth, dentals, head and neck region;
11. Facial psoriasis, eczema, acne, rosacea, perioral dermatitis and herpes zoster in the treatment area;
12. Cancer or precancer in the treatment area, e.g. actinic keratosis;
13. History of bleeding disorders or treatment with thrombolytics, anticoagulants, or inhibitors of platelet aggregation (e.g. Aspirin or other non-steroid anti-inflammatory drugs [NSAIDs]), within 2 weeks before treatment;
14. Patients using immunosuppressants;
15. Patients with a tendency to form hypertrophic scars or any other healing disorders;
16. Patients with known hypersensitivity to lidocaine or agents structurally related to amide type local anaesthetics (e.g., certain anti-arrhythmics);
17. Patients administered dental block or topical administration of lidocaine;
18. Patients with epilepsy, impaired cardiac conduction, severely impaired hepatic function or severe renal dysfunction.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Skin lifting capacity of two Restylane products, as assessed by ultrasound | Baseline
  The lifting capacity of two Restylane products (i.e., Restylane + Lidocaine and Restylane Lyft) will be assessed post-injection, using a skin ultrasound.

SECONDARY OUTCOMES:
Skin lifting capacity of two Restylane products, as assessed by ultrasouns | Week 2
  The lifting capacity of two Restylane products (i.e., Restylane + Lidocaine and Restylane Lyft) will be assessed post-injection, using a skin ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Erevna Innovations Inc, Montreal, Quebec, Canada